CLINICAL TRIAL: NCT04947579
Title: A Phase 2 Multicenter, Randomized, Double-Blinded, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of CC-99677 in Subjects With Active Ankylosing Spondylitis
Brief Title: A Study of CC-99677 in Participants With Active Ankylosing Spondylitis
Acronym: AS SpA axSpA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has been terminated due to Non-Safety reasons because of lack of efficacy in the short-term acute phase.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-99677-AS-001; U1111-1265-3951 (Registry Identifier: UTN Number); 2019-004108-37 (EudraCT Number)
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Spondylitis, Ankylosing
Keywords: Ankylosing Spondylitis; CC-99677; MK2inhibitor; Spinal Diseases; Bone Diseases; Musculoskeletal Diseases; Arthritis; Joint Diseases
MeSH Terms: conditions — Spondylitis, Ankylosing; Spinal Diseases; Bone Diseases; Musculoskeletal Diseases; Arthritis; Joint Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Administration of CC-99677 150 mg QD PO (Experimental): 49 participants will be randomized to CC-99677 150 mg in biologic naive main study
  Interventions: Drug: CC-99677
- Administration of CC-99677 60mg QD PO (Experimental): 49 participants will be randomized to CC-99677 60 mg in biologic naive main study
  Interventions: Drug: CC-99677
- Administration of Placebo QD PO (Placebo Comparator): 49 participants will be randomized to placebo in biologic naive main study
  Interventions: Other: Placebo
- Administration of CC-99677 150 mg QD PO. (Experimental): 20 participants will be randomized to CC-99677 150 mg in biologic-failure substudy
  Interventions: Drug: CC-99677
- Administration of CC-99677 60mg QD PO. (Experimental): 20 participants will be randomized to CC-99677 60 mg in biologic-failure substudy
  Interventions: Drug: CC-99677
- Placebo additional dose cohort (Placebo Comparator): 10 participants will be randomized to placebo in biologic-failure substudy
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CC-99677 — Oral
  Arms: Administration of CC-99677 150 mg QD PO; Administration of CC-99677 150 mg QD PO.; Administration of CC-99677 60mg QD PO; Administration of CC-99677 60mg QD PO.
Other: Placebo — Oral
  Arms: Administration of Placebo QD PO; Placebo additional dose cohort

SUMMARY:
This study is designed to learn about response to CC-99677 treatment by measuring signs and symptoms of Ankylosing Spondylitis (AS), objective measures of disease activity, quality of life assessments, pharmacokinetics, safety, and tolerability over a 12-week double-blind period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ankylosing Spondylitis (AS) fulfilling the modified New York criteria
* Active axial disease at Screening and Baseline defined by a Bath Ankylosing
* Spondylitis Disease Activity Index (BASDAI) score ≥ 4 and Total Back Pain ≥ 4
* Failed prior treatment with at least 2 NSAIDs for at least 4 weeks each
* Participant has never received a biologic therapy eg, tumor necrosis factor (TNF) antagonist or monoclonal antibody [mAb] against IL-17A (biologic naive main study), or have taken more than one biologic therapy (biologic-failure substudy) for the treatment of AS

Exclusion Criteria:

* Radiographic evidence of total ankylosis of the spine
* Clinically significant back pain caused by diseases other than AS
* Concurrent treatment or treatment within the 6 months prior to Baseline with cell depleting biologic agents
* Participation in any study of an investigational drug, including those for COVID-19
* History of malignancy
* Oral corticosteroids (prednisone or equivalent) > 10 mg/day systemically for ≥ 2 weeks prior to Baseline Visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, MD, Study Director — Bristol-Myers Squibb
Locations (63):
- United States (16):
  - Local Institution - 024, Flagstaff, Arizona
  - Local Institution - 021, Gilbert, Arizona
  - Local Institution - 022, Phoenix, Arizona
  - Local Institution - 025, Tucson, Arizona
  - Local Institution - 017, Tustin, California
  - Local Institution - 026, Saint Clair Shores, Michigan
  - Local Institution - 028, Cleveland, Ohio
  - Local Institution - 004, Dayton, Ohio
  - Local Institution - 009, Portland, Oregon
  - Local Institution - 003, Duncansville, Pennsylvania
  - Local Institution - 005, Jackson, Tennessee
  - Local Institution - 002, Memphis, Tennessee
  - Local Institution - 029, Austin, Texas
  - Local Institution - 006, Colleyville, Texas
  - Local Institution - 019, Fort Worth, Texas
  - Local Institution - 008, Houston, Texas
- China (5):
  - Local Institution - 154, Shanghai, Shanghai Municipality
  - Local Institution - 151, Guangzhou
  - Local Institution - 152, Hangzhou
  - Local Institution - 153, Huangpu District
  - Local Institution - 150, Wuhan
- Czechia (8):
  - Local Institution - 205, Brno
  - Local Institution - 206, Ostrava
  - Local Institution - 207, Ostrava
  - Local Institution - 201, Pardubice
  - Local Institution - 202, Prague
  - Local Institution - 203, Prague
  - Local Institution - 211, Prague
  - Local Institution - 204, Uherské Hradište
- Local Institution - 900, Herne, Germany
- Poland (14):
  - Local Institution - 311, Bialystok
  - Local Institution - 315, Bialystok
  - Local Institution - 305, Bydgoszcz
  - Local Institution - 302, Bydgoszcz
  - Local Institution - 301, Elblag
  - Local Institution - 307, Katowice
  - Local Institution - 300, Krakow
  - Local Institution - 308, Krakow
  - Local Institution - 310, Nowa Sól
  - Local Institution - 313, Onyksowa 10
  - Local Institution - 312, Sochaczew
  - Local Institution - 306, Torun
  - Local Institution - 303, Warsaw
  - Local Institution - 309, Wroclaw
- Romania (4):
  - Local Institution - 400, Brasov
  - Local Institution - 404, Bucharest
  - Local Institution - 402, Bucharest
  - Local Institution - 403, Bucharest
- Spain (7):
  - Local Institution - 604, A Coruña
  - Local Institution - 607, Barcelona
  - Local Institution - 606, Córdoba
  - Local Institution - 605, Mérida
  - Local Institution - 601, Sabadell
  - Local Institution - 602, Santiago de Compostela
  - Local Institution - 603, Seville
- Turkey (Türkiye) (8):
  - Local Institution - 702, Adapazarı
  - Local Institution - 707, Altındağ/Ankara
  - Local Institution - 700, Ankara
  - Local Institution - 701, Edirne
  - Local Institution - 705, Istanbul
  - Local Institution - 706, Izmir
  - Local Institution - 704, Karabağlar
  - Local Institution - 703, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants originally randomized to the CC-99677 60 mg or 150 mg Biologic Naive or Biologic Failure arms in the Placebo-Controlled period continued receiving the same intervention until week 64 in the Long-Term Extension period.
Groups:
- Placebo Biologic Naive: Placebo Biologic Naive QD PO from week 0 - 12. At week 12, participants rerandomized to CC-99677 (150 mg or 60 mg PO QD) through Week 64 or until early discontinuation
- CC-99677 60 mg Biologic Naive: CC-99677 60 mg Biologic Naive QD PO through Week 64 or until early discontinuation
- CC-99677 150 mg Biologic Naive: CC-99677 150 mg Biologic Naive QD PO through Week 64 or until early discontinuation
- Placebo Biologic Failure: Placebo Biologic Failure QD PO from week 0 - 12. At week 12, participants rerandomized to CC-99677 (150 mg or 60 mg PO QD) through Week 64 or until early discontinuation
- CC-99677 60 mg Biologic Failure: CC-99677 60 mg Biologic Failure QD PO through Week 64 or until early discontinuation
- CC-99677 150 mg Biologic Failure: CC-99677 150 mg Biologic Failure QD PO through Week 64 or until early discontinuation
Period: Week 0 - Week 12 (Placebo-Controlled)
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Started | 49 | 49 | 49 | 5 | 7 | 8
Completed | 42 | 42 | 39 | 3 | 5 | 7
Not Completed | 7 | 7 | 10 | 2 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other reasons | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 2 | 0
Not completed — Study terminated by sponsor | 5 | 6 | 7 | 1 | 0 | 1
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0 | 0
Period: Week 12 - Week 64 (Long-Term Extension)
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Started | 0 | 63 | 61 (1 participant discontinued in the Placebo-Controlled period but entered the Long-Term Extension period.) | 0 | 7 | 8
Placebo Patients Re-randomized to CC-99677 60 mg | 0 | 21 | 0 | 0 | 2 | 0
Placebo Patients Re-randomized to CC-99677 150 mg | 0 | 0 | 21 | 0 | 0 | 1
Completed | 0 | 1 | 1 | 0 | 0 | 0
Not Completed | 0 | 62 | 60 | 0 | 7 | 8
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 54 | 46 | 0 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 4 | 0 | 1 | 3
Not completed — Other reasons | 0 | 5 | 8 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure | Total
Number analyzed (Participants) | 49 | 49 | 49 | 5 | 7 | 8 | 167
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (10.27) | 40.5 (11.78) | 40.4 (9.75) | 43.8 (7.16) | 44.4 (10.06) | 42.5 (9.46) | 41.9 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 12 | 1 | 1 | 0 | 28
  Male | 41 | 43 | 37 | 4 | 6 | 8 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 47 | 47 | 49 | 5 | 7 | 8 | 163
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 48 | 48 | 48 | 5 | 7 | 8 | 164
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve ASAS 20 at Week 12
Description: Percentage of participants who achieve an improvement in disease activity from baseline of ≥ 20% and ≥ 1 unit in at least 3 of the 4 SpondyloArthritis International Society (ASAS) domains on a scale of 0 to 10, and no worsening from baseline of ≥ 20% and ≥ 1 unit in the remaining domain on a scale of 0 to 10. Baseline is the last non-missing value on or before the date of the first dose of investigational product. The four ASAS Domains are:
  * Patient Global Assessment of Disease (0 to 10 unit Numerical Rating Scale [NRS]);
  * Total Back Pain NRS;
  * Function (the Bath Ankylosing Spondylitis Functional Index [BASFI] score NRS);
  * Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] NRS Questions #5 and #6 for morning stiffness).
Time Frame: Week 12
Population: All treated participants who have non-missing response at week 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Number analyzed (Participants) | 41 | 43 | 41 | 3 | 6 | 7
Percentage of Participants | 48.8 | 51.2 | 56.1 | 66.7 | 83.3 | 57.1
Statistical Analysis 1: Comparison: Placebo Biologic Naive vs CC-99677 60 mg Biologic Naive; Test type: Superiority; p = 0.829, Cochran-Mantel-Haenszel; Stratified difference = 2.4, 95% CI 2-sided [-18.2 to 22.7] — CC99677 60 mg - Placebo
Statistical Analysis 2: Comparison: Placebo Biologic Naive vs CC-99677 150 mg Biologic Naive; Test type: Superiority; p = 0.512, Cochran-Mantel-Haenszel; Stratified difference = 7.3, 95% CI 2-sided [-13.8 to 27.5] — CC99677 150 mg - Placebo

2. Secondary Outcome: Percentage of Participants Who Achieve ASAS 40 at Week 12
Description: Percentage of participants who achieve an improvement in disease activity from baseline of ≥ 40% and ≥ 2 unit in at least 3 of the 4 SpondyloArthritis International Society (ASAS) domains on a scale of 0 to 10, and no worsening at all from baseline in the remaining domain. Baseline is the last non-missing value on or before the date of the first dose of investigational product. The four ASAS Domains are:
  * Patient Global Assessment of Disease (0 to 10 unit Numerical Rating Scale [NRS]);
  * Total Back Pain NRS;
  * Function (the Bath Ankylosing Spondylitis Functional Index [BASFI] score NRS);
  * Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] NRS Questions #5 and #6 for morning stiffness).
Time Frame: Week 12
Population: All treated participants who have non-missing response at week 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Number analyzed (Participants) | 41 | 43 | 41 | 3 | 6 | 7
Percentage of Participants | 22.0 | 25.6 | 34.1 | 33.3 | 50.0 | 28.6
Statistical Analysis 1: Comparison: Placebo Biologic Naive vs CC-99677 60 mg Biologic Naive; Test type: Superiority; p = 0.725, Cochran-Mantel-Haenszel; Stratified difference = 3.3, 95% CI 2-sided [-14.9 to 21.0] — CC99677 60 mg - Placebo
Statistical Analysis 2: Comparison: Placebo Biologic Naive vs CC-99677 150 mg Biologic Naive; Test type: Superiority; p = 0.219, Cochran-Mantel-Haenszel; Stratfied difference = 12.2, 95% CI 2-sided [-7.2 to 30.5] — CC99677 150 mg - Placebo

3. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score With CRP (ASDAS-CRP) at Week 12
Description: ASDAS-CRP is a score of disease activity that combines patient reported assessments of back pain (Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] question 2), duration of morning stiffness (BASDAI question 6), peripheral joint pain and/or swelling (BASDAI question 3), general wellbeing, and CRP in a weighted manner. The cut-off values for disease activity states and improvement scores are defined as follows: <1.3 inactive disease, ≥1.3 and <2.1 low disease activity, ≥2.1 and ≤3.5 high disease activity and 3.5 very high disease activity. The minimum clinically important difference (MCID) are defined as: change of at least 1.1 unit for 'clinically important improvement' and change of at least 2.0 units for 'major improvement'. Baseline is the last non-missing value on or before the date of the first dose of investigational product. ASDAS-CRP Formula: 0.12xBack Pain+0.06xDuration of Morning Stiffness+0.11xPatient Global+0.07xPeripheral Pain/Swelling+0.58xln(CRP+1)
Time Frame: Baseline and Week 12
Population: All treated participants with baseline and week 12 measurements
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Number analyzed (Participants) | 40 | 43 | 41 | 3 | 5 | 7
Units on a scale | -0.69 (0.856) | -0.87 (0.681) | -0.80 (0.869) | -0.84 (0.621) | -1.02 (0.464) | -0.44 (0.323)
Statistical Analysis 1: Comparison: Placebo Biologic Naive vs CC-99677 60 mg Biologic Naive; Test type: Superiority; p = 0.299, Longitudinal data analysis model; Difference in Adjusted Means = -0.17, 95% CI 2-sided [-0.50 to 0.16], Standard Error of Mean 0.167 — CC99677 60 mg - Placebo
Statistical Analysis 2: Comparison: Placebo Biologic Naive vs CC-99677 150 mg Biologic Naive; Test type: Superiority; p = 0.488, Longitudinal data analysis model; Difference in Adjusted Means = -0.12, 95% CI 2-sided [-0.45 to 0.22], Standard Error of Mean 0.168 — CC99677 150 mg - Placebo

4. Secondary Outcome: Change From Baseline in BASDAI at Week 12
Description: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is a composite score based on a self-administered survey of six questions using a 0 to 10 unit numerical rating scale (NRS) that assesses five major symptoms of AS during the last week: 1) fatigue; 2) spinal pain; 3) peripheral joint pain/swelling; 4) areas of localized tenderness; 5a) morning stiffness severity upon wakening; 5b) morning stiffness duration upon wakening. To give each of the five symptoms equal weighting, the mean of the two scores relating to morning stiffness is taken. The resulting 0 to 50 score is divided by 5 to give a final 0 to 10 BASDAI score. A BASDAI score of 4 or greater is considered to be indicative of active AS disease. Baseline is the last non-missing value on or before the date of the first dose of investigational product.
Time Frame: Baseline and Week 12
Population: All treated participants with baseline and week 12 measurements
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Number analyzed (Participants) | 43 | 43 | 41 | 3 | 6 | 7
Units on a scale | -1.88 (1.862) | -1.96 (1.494) | -2.03 (2.080) | -1.63 (0.651) | -2.20 (1.394) | -1.43 (1.517)
Statistical Analysis 1: Comparison: Placebo Biologic Naive vs CC-99677 60 mg Biologic Naive; Test type: Superiority; p = 0.970, Longitudinal data analysis model; Difference in Adjusted Means = 0.01, 95% CI 2-sided [-0.76 to 0.79], Standard Error of Mean 0.391 — CC99677 60 mg - Placebo
Statistical Analysis 2: Comparison: Placebo Biologic Naive vs CC-99677 150 mg Biologic Naive; Test type: Superiority; p = 0.668, Longitudinal data analysis model; Difference in Adjusted Means = -0.17, 95% CI 2-sided [-0.95 to 0.61], Standard Error of Mean 0.393 — CC99677 150 mg - Placebo

5. Secondary Outcome: Change From Baseline in BASFI at Week 12
Description: Bath Ankylosing Spondylitis Functional Index (BASFI) is a composite score based on a self administered survey of ten questions using a 0 to 10 unit numerical rating scale (NRS) that assesses degree of mobility and functional ability during the last week. The questionnaire consists of eight questions regarding function in AS and the two last questions reflecting ability to cope with everyday life. The left-hand box of 0 represents "easy," and the right-hand box represents "impossible." The resulting 0 to 100 score is divided by 10 to give a final 0 to 10 BASFI score. A higher BASFI score correlates to reduced functional ability. Baseline is the last non-missing value on or before the date of the first dose of investigational product.
Time Frame: Baseline and Week 12
Population: All treated participants with baseline and week 12 measurements
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Number analyzed (Participants) | 41 | 43 | 41 | 3 | 6 | 7
Units on a scale | -1.22 (1.727) | -1.33 (1.985) | -1.28 (2.542) | -1.77 (0.850) | -1.47 (1.841) | -1.29 (0.703)
Statistical Analysis 1: Comparison: Placebo Biologic Naive vs CC-99677 60 mg Biologic Naive; Test type: Superiority; p = 0.890, Longitudinal data analysis model; Difference in Adjusted Means = 0.06, 95% CI 2-sided [-0.77 to 0.88], Standard Error of Mean 0.416 — CC99677 60 mg - Placebo
Statistical Analysis 2: Comparison: Placebo Biologic Naive vs CC-99677 150 mg Biologic Naive; Test type: Superiority; p = 0.545, Longitudinal data analysis model; Difference in Adjusted Means = 0.25, 95% CI 2-sided [-0.57 to 1.08], Standard Error of Mean 0.417 — CC99677 150 mg - Placebo

6. Secondary Outcome: Change From Baseline in the SPARCC SI Joint Score at Week 12
Description: Change from Baseline in the Spondyloarthritis Research Consortium of Canada (SPARCC) scores of the sacroiliac joints. The SPARCC assesses 16 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include Medial epicondyle (left/right [L/R]), Lateral epicondyle (L/R), Supraspinatus insertion into greater tuberosity of humerus (L/R), Greater trochanter (L/R), Quadriceps insertion into superior border of patella (L/R), Patellar ligament insertion into inferior pole of patella or tibial tubercle (L/R), Achilles tendon insertion into calcaneum (L/R), and Plantar fascia insertion into calcaneum (L/R). The SPARCC is the sum of all site scores (range 0 to 16). Higher scores indicate more severe enthesitis. Baseline is the last non-missing value on or before the date of the first dose of investigational product.
Time Frame: Baseline and Week 12
Population: All treated participants with baseline and week 12 measurements
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Number analyzed (Participants) | 38 | 43 | 39 | 3 | 5 | 7
Units on a scale | 0.25 (3.168) | -0.81 (5.453) | -1.72 (6.084) | -0.17 (1.258) | -3.00 (7.608) | -3.00 (4.093)
Statistical Analysis 1: Comparison: Placebo Biologic Naive vs CC-99677 60 mg Biologic Naive; Test type: Superiority; p = 0.778, Longitudinal data analysis model; Difference in Adjusted Means = -0.28, 95% CI 2-sided [-2.26 to 1.70], Standard Error of Mean 0.999 — CC99677 60 mg - Placebo
Statistical Analysis 2: Comparison: Placebo Biologic Naive vs CC-99677 150 mg Biologic Naive; Test type: Superiority; p = 0.330, Longitudinal data analysis model; Difference in Adjusted Means = -1.00, 95% CI 2-sided [-3.02 to 1.03], Standard Error of Mean 1.022 — CC99677 150 mg - Placebo

7. Secondary Outcome: Change From Baseline in the SPARCC Spine Score at Week 12
Description: Change from Baseline in the Spondyloarthritis Research Consortium of Canada (SPARCC) scores of the total spine. All 23 disco-vertebral units (DVU) of the spine (from C2 to S1) were scored for bone marrow edema. A single DVU has 18 scoring units, and each has score of 0 or 1, bringing the maximum total score to 414, the sum ranges from 0 to 414 with higher scores reflecting worse disease.
  Baseline is the last non-missing value on or before the date of the first dose of investigational product.
Time Frame: Baseline and Week 12
Population: All treated participants with baseline and week 12 measurements
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Number analyzed (Participants) | 38 | 43 | 39 | 3 | 5 | 7
Units on a scale | -0.92 (7.557) | -1.53 (8.331) | -1.86 (7.081) | -8.17 (7.371) | -2.40 (5.128) | -2.71 (8.640)
Statistical Analysis 1: Comparison: Placebo Biologic Naive vs CC-99677 60 mg Biologic Naive; Test type: Superiority; p = 0.600, Longitudinal data analysis model; Difference in Adjusted Means = -0.82, 95% CI 2-sided [-3.93 to 2.28], Standard Error of Mean 1.567 — CC99677 60 mg - Placebo
Statistical Analysis 2: Comparison: Placebo Biologic Naive vs CC-99677 150 mg Biologic Naive; Test type: Superiority; p = 0.416, Longitudinal data analysis model; Difference in Adjusted Means = -1.31, 95% CI 2-sided [-4.49 to 1.87], Standard Error of Mean 1.605 — CC99677 150 mg - Placebo

8. Secondary Outcome: Percent Change From Baseline in hsCRP at Week 12
Description: Percent change from baseline in high-sensitivity C-reactive protein (hsCRP). Baseline is the last non-missing value on or before the date of the first dose of investigational product.
Time Frame: Baseline and Week 12
Population: All treated participants with baseline and week 12 measurements
Measure: Mean (Standard Deviation); unit: Percent change in hsCRP
Arm/Group | Placebo Biologic Naive | CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Naive | Placebo Biologic Failure | CC-99677 60 mg Biologic Failure | CC-99677 150 mg Biologic Failure
Number analyzed (Participants) | 42 | 43 | 41 | 3 | 5 | 7
Percent change in hsCRP | 72.83 (474.199) | -1.43 (64.157) | 20.88 (130.181) | -13.68 (55.618) | 8.52 (66.057) | 452.34 (1226.664)
Statistical Analysis 1: Comparison: Placebo Biologic Naive; Test type: Superiority; Adjusted Mean = -6.26, 95% CI [-27.31 to 14.79], Standard Error of Mean 10.741
Statistical Analysis 2: Comparison: CC-99677 60 mg Biologic Naive; Test type: Superiority; Adjusted Mean = -18.58, 95% CI 2-sided [-36.57 to -0.58], Standard Error of Mean 9.181
Statistical Analysis 3: Comparison: CC-99677 150 mg Biologic Naive; Test type: Superiority; Adjusted Mean = -12.16, 95% CI 2-sided [-31.96 to 7.65], Standard Error of Mean 10.105

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (Up to approximately 17 months). SAEs and Other AEs were assessed from first dose up to 28 days post last dose (Up to approximately 16 months).
Description: Placebo patients from week 0 - week 12 are reported separately in Biologic Naive or Biologic Failure arms. Placebo patients who are rerandomized at week 12 to CC99677 60 mg or 150 mg are reported separately in "Placebo to CC-99677" Biologic Naive or Biologic Failure arms.
Groups:
- Placebo Biologic Naive: Placebo Biologic Naive QD PO from week 0 - 12
- Placebo to CC-99677 150 mg Biologic Naive; Placebo to CC-99677 150 mg Biologic Failure: At week 12, participants rerandomized to CC-99677 150 mg PO QD through Week 64 or until early discontinuation
- Placebo to CC-99677 60 mg Biologic Naive; Placebo to CC-99677 60 mg Biologic Failure: At week 12, participants rerandomized to CC-99677 60 mg PO QD through Week 64 or until early discontinuation
- Placebo Biologic Failure: Placebo Biologic Failure QD PO from week 0 - 12
Arm/Group | CC-99677 150 mg Biologic Naive | CC-99677 60 mg Biologic Naive | Placebo Biologic Naive | Placebo to CC-99677 150 mg Biologic Naive | Placebo to CC-99677 60 mg Biologic Naive | CC-99677 150 mg Biologic Failure | CC-99677 60 mg Biologic Failure | Placebo Biologic Failure | Placebo to CC-99677 150 mg Biologic Failure | Placebo to CC-99677 60 mg Biologic Failure
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/7 | 1/21 | 0/21 | 0/8 | 0/7 | 0/2 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 1/7 | 3/21 | 0/21 | 3/8 | 0/7 | 1/2 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 11/49 | 26/49 | 0/7 | 8/21 | 7/21 | 6/8 | 4/7 | 1/2 | 1/1 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-99677 150 mg Biologic Naive (N=49) | CC-99677 60 mg Biologic Naive (N=49) | Placebo Biologic Naive (N=7) | Placebo to CC-99677 150 mg Biologic Naive (N=21) | Placebo to CC-99677 60 mg Biologic Naive (N=21) | CC-99677 150 mg Biologic Failure (N=8) | CC-99677 60 mg Biologic Failure (N=7) | Placebo Biologic Failure (N=2) | Placebo to CC-99677 150 mg Biologic Failure (N=1) | Placebo to CC-99677 60 mg Biologic Failure (N=2)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC-99677 150 mg Biologic Naive (N=49) | CC-99677 60 mg Biologic Naive (N=49) | Placebo Biologic Naive (N=7) | Placebo to CC-99677 150 mg Biologic Naive (N=21) | Placebo to CC-99677 60 mg Biologic Naive (N=21) | CC-99677 150 mg Biologic Failure (N=8) | CC-99677 60 mg Biologic Failure (N=7) | Placebo Biologic Failure (N=2) | Placebo to CC-99677 150 mg Biologic Failure (N=1) | Placebo to CC-99677 60 mg Biologic Failure (N=2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 8 | 0 | 1 | 4 | 2 | 0 | 0 | 1 | 0
Genital candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 6 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT04947579/Prot_SAP_000.pdf